CLINICAL TRIAL: NCT06924697
Title: Effect of Glucagon-like Peptide-1 (GLP-1) Receptor Agonist Stimulation on Smoking Consumption in Type 2 Diabetes Patients: Study Protocol of a Randomized, Parallel -Controlled Clinical Trial
Brief Title: Effect of Glucagon-like Peptide-1 (GLP-1) Receptor Agonist Stimulation on Smoking Consumption in Type 2 Diabetes Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC.D(BG).025.04.0
Record Dates: First submitted 2025-03-16; First posted 2025-04-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Nicotine Dependence, Cigarettes
Keywords: clinical pharmacology; functional magnetic resonance imaging; smoking cessation; Diabetes Mellitus, Type 2; GLP-1 receptor agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 group (Experimental)
  Interventions: Drug: Application of GLP-1RAs drugs
- DPP-4i group (Active Comparator)
  Interventions: Drug: DPP-4i group

INTERVENTIONS:
Drug: Application of GLP-1RAs drugs — The pharmacological intervention will be given as an add-on to the standardised psychosocial T2DM treatment paradigm. Patients self-inject Semaglutide once a week or use other GLP-1RAs
  Arms: GLP-1 group
Drug: DPP-4i group — The pharmacological intervention will be given as an add-on to the standardised psychosocial T2DM treatment paradigm. Patients took the DPP-4i according to their actual needs.
  Arms: DPP-4i group

SUMMARY:
Diabetes has become an increasingly serious global health issue. In 2024, approximately 537 million adults were living with diabetes, and this number is projected to rise to 783 million by 2045, representing a 46% increase. Against the backdrop of a growing global diabetes epidemic, smoking among individuals with diabetes poses a significant threat, further exacerbating clinical and public health burdens. Despite over 50 years of tobacco control efforts, smoking remains one of the greatest public health threats in history, causing more than 8 million deaths annually worldwide. Among these, over 7 million deaths result from direct tobacco use, while approximately 1.3 million deaths are attributed to secondhand smoke exposure.

Recent studies have shown that smoking increases the risk of developing prediabetes and diabetes. Moreover, individuals with diabetes who smoke have a higher risk of all-cause mortality, worsened chronic diabetic complications, an increased likelihood of developing cancer and cardiovascular diseases, and greater difficulty in glycemic control. Despite substantial evidence highlighting the detrimental effects of smoking on individuals with diabetes, national surveys from the 1990s indicated similar smoking prevalence rates between individuals with and without diabetes (27.3% and 25.9%, respectively). Although various smoking cessation methods are available, the success rate of quitting remains low, necessitating novel intervention strategies.

Glucagon-like peptide-1 receptor agonists (GLP-1RAs) are widely used in the treatment of type 2 diabetes. They exert hypoglycemic effects by stimulating insulin secretion in a glucose-dependent manner, inhibiting glucagon secretion, enhancing glucose uptake in muscle and adipose tissue, suppressing hepatic glucose production, delaying gastric emptying, and reducing appetite. Existing studies suggest that GLP-1 influences the brain's reward system, and GLP-1RAs have been shown to reduce nicotine dependence in animal models. Recent clinical research has demonstrated that GLP-1RAs can be used in combination with nicotine patches to facilitate smoking cessation. However, whether GLP-1RAs alone can directly promote smoking cessation in individuals with diabetes remains unclear. Therefore, this study aims to investigate the potential direct effects of GLP-1RAs on smoking cessation in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes has become an increasingly severe global health concern. In 2021, an estimated 537 million adults worldwide were living with diabetes, and this number is projected to rise to 783 million by 2045, reflecting a 46% increase. Against the backdrop of the rising global prevalence of diabetes, smoking has been identified as a major risk factor for its onset, as well as a contributor to poor glycemic control and the progression of chronic diabetes complications. Moreover, smoking is an independent risk factor for elevated HbA1c levels. It has been reported that for every additional 20 pack-years of smoking, HbA1c increases by 0.12%. A meta-analysis of 46 prospective studies revealed that smoking increases the risk of all-cause mortality in patients with diabetes by 48%, the risk of coronary heart disease by 54%, myocardial infarction by 52%, and stroke by 44%. Additionally, smoking has been linked to an increased incidence of proteinuria and diabetic nephropathy.

Despite over 50 years of global tobacco control efforts, smoking remains one of the greatest public health threats in history. Tobacco use is responsible for approximately 8 million deaths annually, with over 7 million attributed to direct smoking and around 1.3 million to second hand smoke exposure. Although numerous smoking cessation interventions are available, the success rate remains suboptimal, highlighting the need for novel strategies. Currently, a combination of pharmacotherapy and counseling is considered the most effective approach for smoking cessation. However, findings from two meta-analyses conducted in 2013 and 2016 suggest that outcomes remain unsatisfactory. The withdrawal symptoms and post-cessation weight gain associated with conventional smoking cessation methods are among the leading causes of relapse.

Patients with T2DM often experience increased hunger. Following smoking cessation, the appetite-suppressing effects of nicotine are diminished, leading to increased food intake. Additionally, smoking cessation may alter gut microbiota, further contributing to weight gain. However, weight gain does not negate the long-term benefits of smoking cessation, which significantly reduces the risk of cardiovascular diseases and all-cause mortality. When exploring novel smoking cessation therapies, it is essential to address both nicotine withdrawal syndrome and the adverse metabolic effects of smoking cessation, such as weight gain, to maximize cessation success rates.

Glucagon-like peptide-1 (GLP-1), a gut hormone, has garnered significant research interest. It is an incretin hormone secreted by intestinal L-cells in response to nutrient intake. GLP-1 acts on the hypothalamus to enhance satiety and reduce food intake while also delaying gastric emptying. GLP-1 receptor agonists (GLP-1RA) are widely used for the treatment of T2DM. They exert glucose-lowering effects by stimulating insulin secretion in a glucose-dependent manner, inhibiting glucagon secretion , increasing glucose uptake in muscle and adipose tissues, suppressing hepatic glucose production, delaying gastric emptying, and reducing appetite.

Furthermore, GLP-1 is implicated in the shared neurobiological mechanisms of addiction via the mesolimbic reward system. Endogenous GLP-1 is produced in the nucleus tractus solitarius (NTS) of the brainstem and acts as a neurotransmitter released in multiple brain regions involved in reward processing. This suggests that GLP-1 may modulate addiction-related behaviours by attenuating neural responses in reward-related brain regions. However, no studies have yet investigated the effects of GLP-1RA on smoking cessation in patients with T2DM. In particular, it remains unclear whether GLP-1RA, at standard therapeutic doses for T2DM, can simultaneously reduce nicotine dependence.

Neuroimaging studies have shown that chronic nicotine use induces cognitive, structural, and functional alterations in the brain. Functional imaging research has identified the insula as a critical region involved in smoking behaviour. A negative correlation has been observed between cortical thickness in insular subregions and nicotine dependence. Additionally, functional imaging studies have demonstrated a positive correlation between nicotine dependence and activation of the anterior and posterior insula in response to smoking-related cues. Recent research has further revealed a negative correlation between nicotine dependence and connectivity between the left and right dorsal and left ventral anterior insula and the superior parietal lobule (SPL), including the left precuneus. The insula has thus been identified as a potential target for nicotine dependence treatment. Moreover, the left praecuneus has been proposed as a neuroimaging biomarker for nicotine addiction, with regional homogeneity (ReHo) values in the right superior frontal gyrus and left praecuneus distinguishing nicotine-dependent individuals.

To date, no studies have investigated nicotine dependence in patients with T2DM. Based on these findings, we hypothesize that GLP-1RA may modulate neural responses in reward-processing regions of the brain, thereby reducing nicotine dependence and cigarette consumption in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 18-75 years.
2. Diagnosis of type 2 diabetes mellitus (T2DM) based on the World Health Organization (WHO) criteria.
3. A history of smoking for at least one year.
4. Fagerström Test for Nicotine Dependence (FTND) score ≥4.
5. Eligible for treatment with glucagon-like peptide-1 receptor agonists (GLP1-RAs) or dipeptidyl peptidase-IV (DPP-IV) inhibitors but have not previously used these medications.
6. Patients who fully understand the study, voluntarily participate, and sign the informed consent form.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes or other specific types of diabetes.
2. Presence of diabetic ketoacidosis or severe diabetic complications.
3. Patients with severe cardiovascular, hepatic, renal, neurological, immune, or hematological diseases.
4. Presence of severe infections, malignancies, recent surgeries, or major trauma.
5. A history of severe recurrent hypoglycemia.
6. Severe gastrointestinal disorders, such as gastroparesis.
7. Poor adherence or inability to attend scheduled follow-up visits.
8. A history of pancreatitis or a high risk of developing pancreatitis.
9. Presence of severe psychiatric disorders, including schizophrenia, paranoid psychosis, bipolar disorder, or intellectual disability.
10. Contraindications to magnetic resonance imaging (MRI), such as metallic implants, pacemakers, or claustrophobia.

    -

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-21 (Estimated); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Fagerstrom Test of Nicotine Dependence (FTND) scores | From enrollment to the end of treatment at 24 weeks.At weeks 0 and 24
  To evaluate smoking behavior and nicotine dependence before and after treatment, the Fagerström Test for Nicotine Dependence (FTND) will be administered at weeks 0, 1, 4, 12, and 24. Patient scores will be recorded.

SECONDARY OUTCOMES:
Functional MRI changes | From enrollment to the end of treatment at 24 weeks.At weeks 0 and 24
  fMRI will be conducted at weeks 0 and 24 to investigate potential treatment effects. Resting-state functional connectivity (rsFC) analysis will be performed to assess time-dependent consistency of blood oxygen level-dependent (BOLD) or perfusion fMRI signal fluctuations between different brain regions in the absence of explicit tasks, providing insights into brain activity. Changes in resting-state functional connectivity, structural connectivity, and brain morphology will be analysed in addiction-related brain regions, including the praecuneus, lingual gyrus, and paracentral lobule. All participants will undergo fMRI scans at baseline and after 24 weeks of treatment.
Laboratory testing | From enrollment to the end of treatment at 24 weeks.At weeks 0, 12, and 24
  Blood samples will be collected at baseline (week 0), week 12, and week 24 for the assessment of complete blood count, liver and kidney function, electrolytes, coagulation profile, HbA1c, lipid profile, thyroid function, proinsulin, insulin, and C-peptide levels. Urine samples will be collected at baseline (week 0), week 12, and the final visit (week 24) for urinalysis, with a particular focus on urinary albumin levels and the albumin-to-creatinine ratio for intergroup comparisons.
Exhaled Carbon Monoxide (CO) Test | From enrollment to the end of treatment at 24 weeks.At weeks 0, 12, and 24
  Exhaled CO levels will be assessed at weeks 0, 12, and 24 to monitor smoking status.
Adverse reactions | From enrollment to the end of treatment at 24 weeks.At weeks 0, 4, 12, and 24
  At baseline (week 0), informed consent will be obtained from all participants. Following medical history collection and eligibility assessment based on inclusion and exclusion criteria, patients will be randomly assigned to either the GLP-1RA group or the DPP-4i group. Any adverse events occurring during the study period will also be documented.
BMI | From enrollment to the end of treatment at 24 weeks.At weeks 0, 4, 12, and 24

CONTACTS AND LOCATIONS:
Overall Officials: jun Song, doctoral degree, Study Director — East Hospital, Tongji University School of Medicine, Shanghai
Locations (1):
- Department of Endocrinology, East Hospital, Tongji University School of Medicine, 150 Jimo Road, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient raw data, statistical analysis programs, and the study protocol.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study concludes, IPD will be available.Data will be available for a period of five years following the completion of the study.
Access Criteria: Eligible researchers must submit a detailed research plan, which will be reviewed by the principal investigator before data access is granted. To ensure data security and formal communication, all data-sharing matters must be arranged via the institutional telephone number +86-21-38804518. After approval, the institution will provide the information to the relevant applicants. Personal email addresses will not be accepted as official contact methods.

REFERENCES:
- [Background] Willenborg J, Menzel W, Vetten HJ, Maiss E. Molecular characterization of two alphacryptovirus dsRNAs isolated from Daucus carota. Arch Virol. 2009;154(3):541-3. doi: 10.1007/s00705-009-0314-z. Epub 2009 Jan 23. No abstract available. PMID 19165417
- [Background] Kondoh H, Takagi S, Nomura K, Okada TS. Transdifferentiation of putative neuronal cells of neural retina into lens: A demonstration by chick-quail chimeric cultures. Wilehm Roux Arch Dev Biol. 1983 Sep;192(5):256-261. doi: 10.1007/BF00848657. PMID 28305512
- [Background] Gomez LA, Patino PJ, Novaira HJ, Morales MM, Condino-Neto A. A single nucleotide polymorphism in the promoter region of theNCF-2 gene. Am J Hematol. 2007 Dec;82(12):1124-5. doi: 10.1002/ajh.21015. No abstract available. PMID 17712795
- [Background] Scanlon TC, Dostal SM, Griswold KE. A high-throughput screen for antibiotic drug discovery. Biotechnol Bioeng. 2014 Feb;111(2):232-43. doi: 10.1002/bit.25019. Epub 2013 Aug 29. PMID 23955804
- [Background] Zhang HB, Scheuring CF, Zhang M, Zhang Y, Wu CC, Dong JJ, Li Y. Construction of BIBAC and BAC libraries from a variety of organisms for advanced genomics research. Nat Protoc. 2012 Feb 16;7(3):479-99. doi: 10.1038/nprot.2011.456. PMID 22343430
- [Background] Gallmeier K, Becker E, Kirsten A, Wolke G, Manuwald O, Meyer H, Magnussen H, Nowak D, Heinrich J. Prediction of new-onset asthma and nasal allergy by skin prick test and RAST in a cohort of adults. Eur Respir J. 2014 Jan;43(1):92-102. doi: 10.1183/09031936.00012813. Epub 2013 Sep 13. PMID 24036244
- [Background] Fernandez Rodriguez R. Language, Science and Globalization in the Eighteenth Century. Ber Wiss. 2023 Mar;46(1):38-53. doi: 10.1002/bewi.202200040. Epub 2023 Mar 6. PMID 36876428
- [Background] Ismail E, Orlando G, Corradini ML, Amerio P, Romani GL, Merla A. Differential diagnosis of Raynaud's phenomenon based on modeling of finger thermoregulation. Physiol Meas. 2014 Apr;35(4):703-16. doi: 10.1088/0967-3334/35/4/703. Epub 2014 Mar 12. PMID 24622281
- [Background] Patinadan PV, Tan-Ho G, Choo PY, Low CX, Ho AHY. 'Food for Life and Palliation (FLiP)': a qualitative study for understanding and empowering dignity and identity for terminally ill patients in Asia. BMJ Open. 2021 Apr 13;11(4):e038914. doi: 10.1136/bmjopen-2020-038914. PMID 33849845
- [Background] Perez H, Tah JHM, Mosavi A. Deep Learning for Detecting Building Defects Using Convolutional Neural Networks. Sensors (Basel). 2019 Aug 15;19(16):3556. doi: 10.3390/s19163556. PMID 31443244
- [Background] Nielsen PA. Mutagenicity studies on complex environmental mixtures: selection of solvent system for extraction. Mutat Res. 1992 Jan-Mar;276(1-2):117-23. doi: 10.1016/0165-1110(92)90060-m. PMID 1370102
- [Background] Tao L, Pereira MA. Quantification of carvone, cineole, perillaldehyde, perillyl alcohol and sobrerol by isocratic high-performance liquid chromatography. J Chromatogr A. 1998 Jan 9;793(1):71-6. doi: 10.1016/s0021-9673(97)00867-4. PMID 9468652
- [Background] Lue NF, Kornberg RD. A possible role for the yeast TATA-element-binding protein in DNA replication. Proc Natl Acad Sci U S A. 1993 Sep 1;90(17):8018-22. doi: 10.1073/pnas.90.17.8018. PMID 8367459
- [Background] Kragh-Hansen U, Donaldson D, Jensen PH. The glycan structure of albumin Redhill, a glycosylated variant of human serum albumin. Biochim Biophys Acta. 2001 Nov 26;1550(1):20-6. doi: 10.1016/s0167-4838(01)00264-3. PMID 11738084
- [Background] Stewart DL, Cook LN, Rabalais GP. Successful use of extracorporeal membrane oxygenation in a newborn with herpes simplex virus pneumonia. Pediatr Infect Dis J. 1993 Feb;12(2):161-2. doi: 10.1097/00006454-199302000-00014. No abstract available. PMID 8426779
- [Background] Calman KC, Mouatt BR. Fluoridation of drinking water. It's safe and it reduces dental decay. BMJ. 1993 Aug 7;307(6900):386. doi: 10.1136/bmj.307.6900.386-c. No abstract available. PMID 8374438
- [Background] Green G, Pool R, Harrison S, Hart GJ, Wilkinson J, Nyanzi S, Whitworth JA. Female control of sexuality: illusion or reality? Use of vaginal products in south west Uganda. Soc Sci Med. 2001 Feb;52(4):585-98. doi: 10.1016/s0277-9536(00)00162-3. PMID 11206655
- [Background] Pan A, Wang Y, Talaei M, Hu FB, Wu T. Relation of active, passive, and quitting smoking with incident type 2 diabetes: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2015 Dec;3(12):958-67. doi: 10.1016/S2213-8587(15)00316-2. Epub 2015 Sep 18. PMID 26388413
- [Background] Ehdaie B, Mason MD, Peters CA, Corbett ST. Transurethral placement of vaginal contraceptive device in a patient with neurogenic bladder: a case report and review of the literature. J Pediatr Urol. 2013 Apr;9(2):e107-10. doi: 10.1016/j.jpurol.2012.11.008. Epub 2012 Dec 6. PMID 23219318
- [Background] Karagiannis DA, Soublis V, Kandarakis A. A case of polypoidal choroidal vasculopathy. Periphery is equally important for such patients. Clin Interv Aging. 2009;4:315-7. doi: 10.2147/cia.s6193. Epub 2009 Jun 29. PMID 19750233
- [Background] Kang YA, Paik H, Zhang SY, Chen JJ, Olson OC, Mitchell CA, Collins A, Swann JW, Warr MR, Fan R, Passegue E. Secretory MPP3 reinforce myeloid differentiation trajectory and amplify myeloid cell production. J Exp Med. 2023 Aug 7;220(8):e20230088. doi: 10.1084/jem.20230088. Epub 2023 Apr 26. PMID 37115584
- [Background] Poku R, Amissah F, Alan JK. PI3K Functions Downstream of Cdc42 to Drive Cancer phenotypes in a Melanoma Cell Line. Small GTPases. 2023 Dec;14(1):1-13. doi: 10.1080/21541248.2023.2202612. PMID 37114375
- [Background] Hanson JA, Hsu FP, Jacob AT, Bota DA, Alexandru D. Antivascular endothelial growth factor antibody for treatment of glioblastoma multiforme. Perm J. 2013 Fall;17(4):68-74. doi: 10.7812/TPP/13-081. PMID 24361023
- [Background] Ogun SA, Tewari R, Otto TD, Howell SA, Knuepfer E, Cunningham DA, Xu Z, Pain A, Holder AA. Targeted disruption of py235ebp-1: invasion of erythrocytes by Plasmodium yoelii using an alternative Py235 erythrocyte binding protein. PLoS Pathog. 2011 Feb;7(2):e1001288. doi: 10.1371/journal.ppat.1001288. Epub 2011 Feb 17. PMID 21379566
- [Background] Hu Y, Zong G, Liu G, Wang M, Rosner B, Pan A, Willett WC, Manson JE, Hu FB, Sun Q. Smoking Cessation, Weight Change, Type 2 Diabetes, and Mortality. N Engl J Med. 2018 Aug 16;379(7):623-632. doi: 10.1056/NEJMoa1803626. PMID 30110591
- [Background] Galcheva SV, Martorana D, Iotova VM, Yotov Y, Neri TM, Street ME. Associations between two single nucleotide polymorphisms of the adiponectin gene, its circulating concentrations and cardiometabolic risk factors in prepubertal children with and without abdominal obesity. J Endocrinol Invest. 2013 Nov;36(10):869-75. doi: 10.3275/8972. Epub 2013 May 22. PMID 23698590
- [Background] Palamar M, Degirmenci C, Ertam I, Yagci A. Ocular response analyser measurements and central corneal thickness in ocular rosacea patients. Int Ophthalmol. 2017 Feb;37(1):7-11. doi: 10.1007/s10792-016-0218-3. Epub 2016 Mar 12. PMID 26971098
- [Background] Clasen FJ, Pierneef RE, Slippers B, Reva O. EuGI: a novel resource for studying genomic islands to facilitate horizontal gene transfer detection in eukaryotes. BMC Genomics. 2018 May 3;19(1):323. doi: 10.1186/s12864-018-4724-8. PMID 29724163
- [Background] Dorum G, Kaur N, Gysi M. Pedigree-based relationship inference from complex DNA mixtures. Int J Legal Med. 2017 May;131(3):629-641. doi: 10.1007/s00414-016-1526-x. Epub 2017 Jan 19. PMID 28101646
- [Background] Wittmann C, Heinzle E. Application of MALDI-TOF MS to lysine-producing Corynebacterium glutamicum: a novel approach for metabolic flux analysis. Eur J Biochem. 2001 Apr;268(8):2441-55. doi: 10.1046/j.1432-1327.2001.02129.x. PMID 11298764
- [Background] Correction to Lancet Diabetes Endocrinol 2022; 10: 741-60. Lancet Diabetes Endocrinol. 2022 Nov;10(11):e11. doi: 10.1016/S2213-8587(22)00280-7. Epub 2022 Oct 7. No abstract available. PMID 36215990